CLINICAL TRIAL: NCT05546970
Title: Efficacy of the Transversus Abdominis Plane Block (TAP-Block) on Analgesia After Cephalic Duodeno-pancreatectomy
Brief Title: Efficacy of the Transversus Abdominis Plane Block on Analgesia After Cephalic Duodeno-pancreatectomy
Acronym: TAP-Block
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8703
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Neoplasms
Keywords: Neoplastic Disease; Pancreatic neoplasia; Pancreatic Neoplasms; Transversus Abdominis Plane Block; TAP-Block; Cephalic duodeno-pancreatectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic duodenectomy is one of the treatments offered to patients with neoplastic disease of the pancreas. In France, in 2018, 14,000 duodeno-pancreatectomies were performed, including 140 at the Hautepierre hospital at the Strasbourg University Hospital. Pancreaticoduodenectomy is a major surgery, causing significant postoperative pain that should be minimized through multimodal analgesia involving in particular locoregional anesthesia. Since 2019, the recommendations of the ERAS company concerning ERAS (Improved Rehabilitation After Surgery) after pancreaticoduodenectomy recommend the establishment of thoracic epidural analgesia in order to limit postoperative pain. When there is a contraindication to the placement of a thoracic epidural, in particular due to arterial and/or venous vascular reconstructions requiring potential perioperative curative anticoagulation, the administration of local anesthetic by pericatricial catheter is recommended. recommended. The Transversus Abdominis Plane (TAP) block has proven analgesic efficacy, safety and harmlessness in colorectal surgery.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years of age)
* Subject operated at HUS for cephalic duodeno-pancreatectomy between 01/01/2018 and 01/04/ 2022.
* Subject who has not expressed an objection to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his/her opposition to participate in the study
* Admission in intensive care unit after the operation
* Morphine treatment at home
* Drug addiction, weaned or not

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years of age) operated at HUS for cephalic duodeno-pancreatectomy between 01/01/2018 and 01/04/ 2022
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of the echo-guided TAP Block on analgesia | Morphine consumption in the first 24 postoperative hours

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie, Réanimation et Médecine péri-Opératoire - CHU de Strasbourg - France, Strasbourg, France